CLINICAL TRIAL: NCT07350018
Title: Comparison of the Efficacy of Calfactant and Poractant Alfa Surfactants Administered by a Less Invasive Surfactant Administration Technique in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Calfactant vs Poractant Alfa Using a Less Invasive Technique in Preterm Infants With Respiratory Distress Syndrome
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Salih Çağrı Çakır, Associate professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-20/9
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Distress Syndrome in Premature Infants; Respiratory Distress Syndrome (RDS); Surfactant
Keywords: Respiratory Distress Syndrome; Premature infant; Poractant alfa; Calfactant; surfactant treatment; Less Invasive Surfactant Administration; LISA
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Respiratory Distress Syndrome; Premature Birth | interventions — poractant alfa; calfactant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Poractant alfa (LISA) (Active Comparator): Preterm infants with respiratory distress syndrome (RDS) will receive poractant alfa via the Less Invasive Surfactant Administration (LISA) technique while on noninvasive respiratory support.
  Interventions: Drug: Poractant alfa
- Calfactant (LISA) (Active Comparator): Preterm infants with respiratory distress syndrome (RDS) will receive calfactant via the Less Invasive Surfactant Administration (LISA) technique while on noninvasive respiratory support.
  Interventions: Drug: Calfactant

INTERVENTIONS:
Drug: Poractant alfa — Poractant alfa will be administered using the Less Invasive Surfactant Administration (LISA) technique. A thin catheter will be inserted into the trachea under direct laryngoscopic visualization, without the need for endotracheal intubation, while the infant continues to breathe spontaneously on noninvasive respiratory support. Dosing and administration will follow standard clinical guidelines. (200 mg/kg initial dose, 100 mg/kg repeat dose)
  Arms: Poractant alfa (LISA)
Drug: Calfactant — Calfactant will be administered using the Less Invasive Surfactant Administration (LISA) technique. A thin catheter will be inserted into the trachea under direct laryngoscopic visualization, without the need for endotracheal intubation, while the infant continues to breathe spontaneously on noninvasive respiratory support. Dosing and administration will follow standard clinical guidelines. (100 mg/kg initial and repeat dose)
  Arms: Calfactant (LISA)

SUMMARY:
Respiratory distress syndrome (RDS) is a common cause of respiratory failure in preterm infants and is frequently treated with surfactant therapy. With the increasing use of noninvasive ventilation, less invasive methods of surfactant administration have been developed. In the technique known as Less Invasive Surfactant Administration (LISA), surfactant is delivered into the trachea through a thin catheter, without the need for endotracheal intubation. This approach may reduce lung injury and improve respiratory outcomes in spontaneously breathing preterm infants. This multicenter, prospective, randomized study aims to compare the clinical effectiveness of poractant alfa and calfactant when administered using the LISA technique in preterm infants born at less than 30 weeks' gestation with RDS who are not intubated. The study will evaluate short-term outcomes, including the need for intubation, repeat surfactant administration, and respiratory support during the first 72 hours of life, as well as longer-term outcomes such as bronchopulmonary dysplasia and other neonatal morbidities.

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) remains one of the leading causes of respiratory failure in preterm infants. Surfactant replacement therapy is a cornerstone of RDS management; however, traditional administration through endotracheal intubation and mechanical ventilation may contribute to ventilator-induced lung injury and increase the risk of adverse pulmonary outcomes. With the widespread adoption of non-invasive respiratory support strategies, less-invasive approaches to surfactant administration have gained increasing attention.

Less Invasive Surfactant Administration (LISA) is a technique in which surfactant is delivered directly into the trachea via a thin catheter under direct laryngoscopic visualization. At the same time, the infant continues to breathe spontaneously on noninvasive respiratory support. This method avoids endotracheal intubation and mechanical ventilation and has been associated with reduced need for invasive ventilation and improved respiratory outcomes in preterm infants.

Several surfactant preparations are currently used in neonatal practice. Poractant alfa and calfactant are two commonly administered natural surfactants with differing biochemical composition and dosing characteristics. Although both agents are widely used for the treatment of RDS, data directly comparing their effectiveness when administered via the LISA technique are limited.

This multicenter, prospective, randomized study is designed to compare the clinical efficacy of poractant alfa and calfactant administered using the LISA technique in preterm infants with respiratory distress syndrome. Eligible participants will be preterm infants born at less than 30 weeks' gestation, diagnosed with RDS based on clinical and radiographic criteria, who are spontaneously breathing and receiving noninvasive respiratory support without prior endotracheal intubation.

After enrollment, infants will be randomly assigned to receive either poractant alfa or calfactant via the LISA method. In both groups, surfactant will be administered through a thin catheter inserted into the trachea under direct laryngoscopic visualization while maintaining spontaneous breathing and noninvasive respiratory support. Standard neonatal intensive care practices will be applied throughout the study period in all participating centers.

The primary focus of the study is to compare short-term respiratory outcomes between the two treatment groups. These include the need for endotracheal intubation, the requirement for repeat surfactant administration, and the level and duration of respiratory support within the first 72 hours of life. Secondary outcomes include longer-term clinical outcomes such as the development of bronchopulmonary dysplasia at 36 weeks' postmenstrual age, as well as other neonatal morbidities, including intraventricular hemorrhage, necrotizing enterocolitis, and overall survival to discharge.

By directly comparing poractant alfa and calfactant administered via the LISA technique in a randomized, multicenter setting, this study aims to provide evidence on the optimal surfactant choice for less invasive treatment of RDS in very preterm infants. The findings are expected to inform clinical practice and contribute to the improvement of respiratory management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Born at a participating study center hospital.
* Gestational age between 24 1/7 and 29 6/7 weeks (<30 0/7 weeks).
* Postnatal age within the first 6 hours of life.
* Being on non-invasive respiratory support.
* Presence of clinical and radiological findings consistent with respiratory distress syndrome (RDS).
* Indication for surfactant therapy defined as a requirement for FiO₂ >30% to achieve target oxygen saturation (SpO₂ 90-94%) while receiving noninvasive respiratory support with a minimum pressure of 6 cmH₂O.
* Written informed consent obtained from a parent or legal guardian.

Exclusion Criteria:

* Infants who were intubated for any reason before the decision to administer surfactant.
* Severe birth asphyxia, defined as the need for advanced resuscitation after birth, 10th minute Apgar score ≤5, and arterial blood gas within the first hour of life showing pH <7.0 and base excess (BE) ≤-12.
* Presence of major congenital anomalies.
* Respiratory distress due to causes other than respiratory distress syndrome (RDS).
* Congenital heart disease.
* Congenital diaphragmatic hernia.
* Pulmonary hypoplasia.
* Chromosomal abnormalities.
* Presence of pneumothorax.
* Lack of informed consent.
* Neonatal seizures presence.
* Postnatal age greater than 6 hours.
* Infants born outside of gestational weeks 24 1/7 - 29 6/7.
* Requirement for invasive mechanical ventilation at enrollment.
* Infants receiving noninvasive respiratory support with an FiO₂ requirement <0.30.

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Need for endotracheal intubation within the first 72 hours of life | Up to 72 hours after birth.
  The need for endotracheal intubation within the first 72 hours of life in preterm infants born at 24 1/7-29 6/7 weeks' gestation receiving calfactant or poractant alfa via LISA.

SECONDARY OUTCOMES:
Need for Repeat Surfactant Administration | Up to 72 hours after birth.
  The requirement for repeat doses of surfactant after the initial LISA procedure in preterm infants treated with calfactant or poractant alfa.
Adverse Events During Surfactant Administration | During the surfactant administration and up to 72 hours after birth.
  The occurrence of adverse events during surfactant administration via LISA, including apnea, bradycardia, oxygen desaturation, surfactant reflux, coughing, laryngospasm, and vomiting.
Bronchopulmonary dysplasia | At 36 weeks' postmenstrual age or discharge, whichever occurred first.
  The incidence of bronchopulmonary dysplasia at 36 weeks' postmenstrual age in preterm infants receiving calfactant or poractant alfa via LISA.
Retinopathy of Prematurity | From birth until discharge, assessed up to 44 weeks' postmenstrual age.
  The incidence of retinopathy of prematurity (ROP) in preterm infants receiving calfactant or poractant alfa via LISA.
Patent Ductus Arteriosus | From birth until the date of the first documented patent ductus arteriosus requiring medical or surgical treatment or the date of hospital discharge, whichever came first, assessed up to 36 weeks' postmenstrual age.
  The incidence of patent ductus arteriosus requiring medical or surgical treatment in preterm infants treated with calfactant or poractant alfa via LISA.
Air Leak Syndromes | Up to 7 days after birth.
  The occurrence of air leak syndromes (including pneumothorax, pulmonary interstitial emphysema, and pneumomediastinum) in preterm infants receiving calfactant or poractant alfa via LISA.
Duration of Respiratory Support | From birth until discontinuation of respiratory support or discharge, whichever occurs first. (Through study completion, an average of 1 year.)
  Total duration of invasive and noninvasive mechanical ventilation.
Length of Hospital Stay | From birth until discharge. (Through study completion, an average of 1 year.)
  Length of hospital stay in days for preterm infants treated with calfactant or poractant alfa via LISA.
Mortality | From the date of randomization until the date of death from any cause or the date of discharge, whichever came first. (Through study completion, an average of 1 year.)
  All-cause mortality before hospital discharge.
Intraventricular Hemorrhage | Up to the 7th day after birth.
  The incidence of intraventricular hemorrhage (IVH) in preterm infants receiving calfactant or poractant alfa via LISA.
Necrotizing Enterocolitis | From birth until the date of the first documented necrotizing enterocolitis or the date of discharge, whichever came first, assessed up to 36 weeks' postmenstrual age.
  The incidence of necrotizing enterocolitis (NEC) in preterm infants receiving calfactant or poractant alfa via LISA.

CONTACTS AND LOCATIONS:
Locations (5):
- Turkey (Türkiye) (5):
  - Bursa City Hospital, Bursa
  - Division of Neonatology, Department of Pediatrics, Bursa Uludağ University Faculty of Medicine, Bursa
  - Division of Neonatology, Department of Pediatrics, University of Health Sciences Bursa Yuksek İhtisas Training and Research Hospital, Bursa
  - Dörtçelik Children's Diseases Hospital, Bursa
  - Medicana Bursa Hospital, Bursa

IPD SHARING:
Plan to Share IPD: No
I am not authorized to share patient data.

REFERENCES:
- [Background] Kakkilaya V, Gautham KS. Should less invasive surfactant administration (LISA) become routine practice in US neonatal units? Pediatr Res. 2023 Apr;93(5):1188-1198. doi: 10.1038/s41390-022-02265-8. Epub 2022 Aug 19. PMID 35986148
- [Background] Sweet DG, Carnielli VP, Greisen G, Hallman M, Klebermass-Schrehof K, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome: 2022 Update. Neonatology. 2023;120(1):3-23. doi: 10.1159/000528914. Epub 2023 Feb 15. PMID 36863329